CLINICAL TRIAL: NCT06686212
Title: Comparative Effects of Sensory Re-education and Neural Mobilization in Carpal Tunnel Syndrome Patients
Brief Title: Comparative Effects of Sensory Re-education and Neural Mobilization in CTS Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0233
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal tunnel syndrome, Grip strength, Sensory reeducation,
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Sensory re-education program, strengthening exercises and kinesio taping (Experimental): The patient will be given a session of 60 minutes 3 days in a week which includes : Splinting (15 minutes), Topical anesthesia spray (10 minutes ) and wrist massage (10 minutes).
  * PNF using upper extremity (D2) pattern (5 minutes).
  * Strengthening exercises (20 minutes) and Kinesio taping for 12 weeks.
  Interventions: Other: Sensory re-education+ strengthening exercises+ kinesio taping
- Group B:Neural mobilization of median nerve, strengthening exercises and kinesio taping. (Experimental): The patient will be given a session of 60 minutes 3 days in a week which includes: ,Median nerve mobilization through various steps of gliding. (30 minutes).
  * Free the bird exercise. (10 minutes).
  * Strengthening exercises (20 minutes) and kinesio taping for 12 weeks.
  Interventions: Other: Neural mobilization+ Strengthening exercises+ Kinesio taping.

INTERVENTIONS:
Other: Sensory re-education+ strengthening exercises+ kinesio taping — Sensory re-education. Splinting: as constant maintained touch with wrist holding in neutral position for 15 minutes.
  Topical anesthesia spray on affected area for 10 minutes. Massage: apply massage over sensitive areas with same speed and pressure, then the light pressure with cotton, velvet, terry cloth, polyester and wool over sensitive area for 10 minutes.
  PNF using upper extremity (D2) pattern including shoulder extension, adduction, internal rotation, wrist and fingers flexed and wrist ulnar deviated. 10-15 repetitions for 5 minutes.
  Strengthening exercises: wrist flexion and extension, supination and pronation, opposition, gripping, ball squeeze and fingers pinching against resistance. 10-15 repetitions of each exercise for 20 minutes.
  Kinesio taping: Taping will be applied twice a week for 12 weeks.
  Arms: Group A: Sensory re-education program, strengthening exercises and kinesio taping
Other: Neural mobilization+ Strengthening exercises+ Kinesio taping. — The median nerve is mobilized through wrist flexion and extension with elbow straight and palm facing up.
  Wrist flexion and extension with elbow flexed to 90 degrees with palm facing up 10-15 repetitions.
  Wrist flexors stretch with extended arm and palm facing down 10-15 repetitions. Straight fist: hold your hand up with fingers straight. Full fist: bend your fingers to form a full fist. Median nerve stretch and wrist extension exercises for 30 minutes. Free the bird exercises, busy bee flexion shape of Z exercises and wall stretch exercise. (10-15 repetitions) for 10 minutes.
  Strengthening exercises: wrist flexion and extension, supination and pronation, opposition, gripping, ball squeeze and fingers pinching against resistance. 10-15 repetitions each for 20 minutes.
  Kinesio taping: The taping will be applied twice a week for 12 weeks.
  Arms: Group B:Neural mobilization of median nerve, strengthening exercises and kinesio taping.

SUMMARY:
The aim of study is to compare the effects of sensory re-education and neural mobilization in CTS patients.

DETAILED DESCRIPTION:
This study will be randomized clinical trial that will be conducted at Services Hospital Lahore and Government Teaching Hospital Shahdara. In this study 48 participants with CTS will be included as per sample size calculation through non-probability convenience sampling technique. Participants that achieve the required standards of inclusion and exclusion criteria will be randomly allocated using online randomization tool into two groups. Group A will receive Sensory Re-education therapy, strengthening exercises and Kinesio taping for 60 minutes, Group B will be given neural mobilization techniques, strengthening exercises and Kinesio taping for 60 minutes with short rest intervals. Both treatments will be given 3 days per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders age 20-50 years with mild and moderate carpal tunnel syndrome.
* Patients having positive score on CTS specific test (Phalen's test and Tinel's test).
* Patients with pain, paresthesia and hyperesthesia at the course of median nerve.
* Patients that are clinically diagnosed with carpal tunnel syndrome by physician. Patients having BMI >25 (kg/m2).

Exclusion Criteria:

* Patients with polyneuropathies.
* Patients with carpal tunnel syndrome due to any systemic illness (diabetes mellitus, thyroid diseases and R.A).

Patients having cervical radiculopathy.

Patients with history of wrist fracture.

Patients getting steroid injections and after CTS surgery.

Obese and pregnant female with carpal tunnel syndrome.

Patients with any cognitive or neurological problems are excluded from study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | 12th week
  The NPRS is use to capture the patient's level of pain. Patients are allowed to indicate the intensity of their current pain level using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).
Boston Carpal Tunnel Questionnaire | 12th week
  A patient self-reported questionnaire includes 2 sub scales: The Symptom Severity Scale (SSS), which comprise 11 questions and uses a 5- point Likert scale; and the Functional Status Scale (FSS) having 8 items, which have to be evaluated for degree of difficulty on a 5-point Likert scale. Each scale generates a final score (sum of scores divided by number of items), which ranges from 1 to 5, with a higher score predicting greater disability.
Hand Held Dynamometer | 12th week
  Hand grip strength is measured using a handheld dynamometer. Patients are asked to grip the dynamometer isometrically and advised to grip it as hard as they can. Readings will be taken in pounds lb. The average value of 3 trials is recorded.
Pinch gauge meter | 12th week
  Tip pinch grip strength will be assessed using a manual dynamometer (pinch gauge meter). Participants asked to perform a maximal pinch grip by pressing the gauge between the tip of their thumb and index finger. The average of three trials will calculated and defined as the maximal tip pinch grip strength measured in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Phd, Study Chair — Riphah International University Lahore Punjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheereen FJ, Sarkar B, Sahay P, Shaphe MA, Alghadir AH, Iqbal A, Ali T, Ahmad F. Comparison of Two Manual Therapy Programs, including Tendon Gliding Exercises as a Common Adjunct, While Managing the Participants with Chronic Carpal Tunnel Syndrome. Pain Res Manag. 2022 Jun 8;2022:1975803. doi: 10.1155/2022/1975803. eCollection 2022. PMID 35719196
- [Background] Jimenez-Del-Barrio S, Cadellans-Arroniz A, Ceballos-Laita L, Estebanez-de-Miguel E, Lopez-de-Celis C, Bueno-Gracia E, Perez-Bellmunt A. The effectiveness of manual therapy on pain, physical function, and nerve conduction studies in carpal tunnel syndrome patients: a systematic review and meta-analysis. Int Orthop. 2022 Feb;46(2):301-312. doi: 10.1007/s00264-021-05272-2. Epub 2021 Dec 3. PMID 34862562
- [Background] Hassan A, Beumer A, Kuijer PPFM, van der Molen HF. Work-relatedness of carpal tunnel syndrome: Systematic review including meta-analysis and GRADE. Health Sci Rep. 2022 Nov 2;5(6):e888. doi: 10.1002/hsr2.888. eCollection 2022 Nov. PMID 36340637
- [Background] Abdolrazaghi HA, Khansari M, Mirshahi M, Ahmadi Pishkuhi M. Effectiveness of Tendon and Nerve Gliding Exercises in the Treatment of Patients With Mild Idiopathic Carpal Tunnel Syndrome: A Randomized Controlled Trial. Hand (N Y). 2023 Mar;18(2):222-229. doi: 10.1177/15589447211006857. Epub 2021 Apr 15. PMID 33855879
- [Background] Lam NW, Goh HT, Kamaruzzaman SB, Chin AV, Poi PJ, Tan MP. Normative data for hand grip strength and key pinch strength, stratified by age and gender for a multiethnic Asian population. Singapore Med J. 2016 Oct;57(10):578-584. doi: 10.11622/smedj.2015164. Epub 2015 Nov 13. PMID 26768064
- [Background] Almasi-Doghaee M, Boostani R, Saeedi M, Ebrahimzadeh S, Moghadam-Ahmadi A, Saeedi-Borujeni MJ. Carpal compression, Phalen's and Tinel's test: Which one is more suitable for carpal tunnel syndrome? Iran J Neurol. 2016 Jul 6;15(3):173-4. No abstract available. PMID 27648179
- [Background] Du J, Yuan Q, Wang XY, Qian JH, An J, Dai Q, Yan XY, Xu B, Luo J, Wang HZ. Manual Therapy and Related Interventions for Carpal Tunnel Syndrome: A Systematic Review and Meta-Analysis. J Integr Complement Med. 2022 Dec;28(12):919-926. doi: 10.1089/jicm.2022.0542. Epub 2022 Jul 27. PMID 35895497
- [Background] Ijaz MJ, Karimi H, Ahmad A, Gillani SA, Anwar N, Chaudhary MA. Comparative Efficacy of Routine Physical Therapy with and without Neuromobilization in the Treatment of Patients with Mild to Moderate Carpal Tunnel Syndrome. Biomed Res Int. 2022 Jun 22;2022:2155765. doi: 10.1155/2022/2155765. eCollection 2022. PMID 35782066